CLINICAL TRIAL: NCT06697587
Title: Enhanced Cognitive Reappraisal and Emotion Awareness Training (eCREAT) for Maladaptive Anger Inhibition - A Pilot Study
Acronym: eCREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hugo Hesser, Professor Hugo Hesser, Örebro University, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230417601
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Maladaptive Anger Inhibition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eCREAT (Experimental): eCREAT consists of four guided internet modules delivered over four weeks (one each week), see "intervention description" below for further details.
  Interventions: Behavioral: Enhanced Cognitive Reappraisal and Emotion Awareness Training (eCREAT)

INTERVENTIONS:
Behavioral: Enhanced Cognitive Reappraisal and Emotion Awareness Training (eCREAT) — eCREAT features psychoeducational content on anger management, practical exercises, and homework assignments, all supported by an online therapist who provides text-based feedback. The protocol builds on a previously evaluated protocol for maladaptive anger (ClinicalTrials.gov; ID: NCT03858296) with added focus on anger inhibition.
  eCREAT is based on the two-stage model of maladaptive anger inhibition (Burns et al., 2008), which posits that suppressed anger may rebound and return as angry fantasies and ruminations. To address these core mechanisms, the treatment includes training on adaptive anger processing and expression and strategies for disrupting anger ruminations. These added treatment components are based on established protocols for depressive rumination, and assertive expression of emotion, adapted for an anger context. Additionally, the treatment also focuses on how to flexibly shift between different emotion regulation strategies depending on contextual demands.

SUMMARY:
Habitual suppression of intense anger, commonly known as maladaptive anger inhibition, is a widespread issue related to various adverse outcomes. These include, for instance, diminished social support, reduced relationship quality, increased risk for coronary heart disease, and heightened susceptibility to chronic and temporary pain conditions. Developing effective psychological treatments may be one key approach to alleviate the distress experienced amongst these individuals.

The overall goal of this pilot study is to further develop and enhance a previously evaluated treatment protocol for maladaptive anger (Bjureberg et al., 2023) to more effectively target maladaptive anger inhibition. The specific goals are:

1. To assess the feasibility and acceptability of the study (operationalized as number of completed modules and measurements, reported negative events and patient experience).
2. To assess outcome variability and estimate the relative effect of the treatment in reducing maladaptive anger inhibition. Maladaptive anger inhibition was operationalized as high levels of trait anger suppression (main outcome), anger rumination (secondary outcome) as well as low levels assertive expression of anger (secondary outcome).

   Secondary aims (to be reported in secondary papers)
3. To assess and explore participants' qualitative experiences of maladaptive anger inhibition.
4. To explore within-subjects emotion dynamics using daily assessments.

DETAILED DESCRIPTION:
1. Treatment feasibility and acceptability will be assessed by measuring treatment retention and adherence (operationalized as number of drop-outs, completed modules, homework assignments, and assessments), treatment credibility and satisfaction (using questionnaires), number of reported adverse events and patient experiences following treatment (see below for details).
2. Following the intention to treat principle data will be analyzed using all participants that were included in the treatment. Preliminary treatment efficacy will be determined by assessing the phase effect of the treatment for each respective outcome (trait anger suppression, anger rumination, and anger assertiveness). More specifically, an interrupted time series design will be used to compare the difference in effect between the treatment phase and a prolonged baseline phase, each consisting of 4 assessments (totaling 8 measurement points). The primary phase effects will be evaluated at treatment termination. Moreover, we will also explore whether treatment effects are maintained at the 3-month follow-up.
3. A subset of 10 consenting participants will be invited to post-treatment interviews. Participants will chosen so as to ensure representation across demographic and clinical variables such as age, gender, and whether they improved or not on the main outcome (trait anger suppression). Interviews will both focus on treatment experiences (goal 1) and participants' qualitative experiences of maladaptive anger inhibition (goal 3).
4. Participants will complete two bursts of 7 days of daily measures of anger and anger regulation strategies, one burst before treatment and one after). These daily measurements will be used to explore within-subject emotion dynamics by comparing emotion dynamics before and after the treatment using dynamic structural equation modeling (DSEM) as our analytical method.

Assessment procedure:

Participants will undergo intensive assessment throughout the project. Participants will complete 1 screening assessment followed by 4 weeks of weekly baseline assessments, with one of the weeks including daily assessments (burst 1). Following the baseline phase, participants will enroll in a 4-week online treatment with weekly assessments. After treatment, participants will undergo 1 week of daily assessments (burst 2) and a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Experience of maladaptive anger inhibition as indicated by a score on the upper quartile on the Anger Expression-In scale from State-Trait Anger Expression Inventory-2 (STAXI-2).

Exclusion Criteria:

* Risk for violence and harm to others.
* Prior convictions of violence/abuse.
* Ongoing psychological treatment.
* Change in psychotropic medication within 2 months prior to enrollment.
* Severe psychiatric disorder, such as severe depression or psychotic disorder
* Ongoing substance use.
* Life circumstances that interfere with treatment.
* Suicidal ideation.
* Not able to read and write in Swedish or learning difficulties (the treatment-format requires normal literacy skills).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger Expression Inventory-2, Anger-Expression In scale (STAXI-2; AX-I) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up.
  Used to assess symptom severity of maladaptive anger inhibition. The AX-I scale has 8 items, each rated on a 4 point, with higher scores reflecting higher degree of anger inhibition. Self-rated.

SECONDARY OUTCOMES:
Behavioral Anger Response Questionnaire, Assertion scale (BARQ; assertion) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up.
  Used to assess the level of assertive expression of anger. The assertion scale has 6 items, each rated on a 5-point scale, with higher scores indicating greater anger assertion. Self-rated.
Anger Rumination Scale (ARS) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up.
  Used to assess levels anger rumination. The scale has 19 items, each rated on a 4-point scale, with higher scores indicating greater levels of anger rumination. Self-rated.
Self-Critical Rumination Scale (SCRS) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up.
  Used to assess levels of self-critical rumination. The scale has 10 items, each rated on a 4-point scale, with higher scores indicating greater levels of self-critical rumination. Self-rated.
Thought Suppression Inventory - Revised, Suppression attempts scale (TSI; Suppression attempts) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up.
  Used to assess levels of thought suppression, adapted for measuring suppression of angry thoughts. The suppression attempts scale has 7 items, each rated on a 5-point scale, with higher scores indicating greater levels of attempts to suppress angry thoughts. Self-rated.
Emotion Regulation Questionnaire (ERQ) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up.
  Used to assess the degree of usage of cognitive reappraisal and expressive suppression, as two emotion regulation strategies. ERQ consists of 10 items divided on two scales that measure cognitive reappraisal (6 items) and expressive suppression (4 items) respectively. Each item is rated on a 7-point scale, with higher scores indicating greater usage of either cognitive reappraisal or expressive suppression. Self-rated.
Five Facets Mindfulness Questionnaire (FFMQ) | Screening, 4 weeks baseline (weekly), 4 weeks treatment (weekly), and 3-month follow-up (see description for details).
  Used to assess the degree of usage of different facets of mindfulness to regulate emotions. FFMQ consists of 29 items and the following scales, each measuring different facets of mindfulness: Observing, Describing, Acting with Awareness, Nonjudging, and Nonreactivity. Each item is rated on a 5-point scale, with higher scores reflecting greater usage of that specific mindfulness facet. Self-rated.
  Additional info about time frame: In this study the Describing and Nonjudging scales were assessed at each assessment point whereas the Acting with Awareness, and Nonreactivity scales were only assessed at screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up. The observing scale was not included in this study.
Aggression Questionnaire (AQ) | Screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up.
  Used to assess level of aggression. AQ consists of 29 items and the following scales: verbal aggression, physical aggression, hostility and anger. For this study we only used the verbal aggression, physical aggression, and hostility scales. Each item is rated on a 4-point scale, with higher score reflecting greater levels of aggression. Self-rated.
Indirect Aggression Scale for perpetrators (IAS-A) | Screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up.
  Used to assess three dimensions of passive aggression. IAS-A consists of 25 items and the following scales: social exclusion, malicious humor and guilt induction. Each item is rated on a 5-point scale, with higher scores representing greater use of passively aggressive behavior. Self-rated.
Perth Alexithymia Questionnaire-Short Form (PAQ-S) | Screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up.
  Used to assess difficulties with identifying and describing emotional experiences (i.e., Alexithymia). PAQ-S consists of 6 items, each item israted on a 7-point scale, with higher scores representing greater problems with Alexithymia. Self-rated.
Difficulties with Emotion Regulation Scale-16 (DERS-16) | Screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up
  Used to assess difficulties with regulating emotions. DERS consists of 16 items and the following scales: clarity, goals, impulse, emotion regulation, and nonacceptance. Each item is rated on a 5-point scale, with higher scores representing greater difficulties with regulating emotions. Self-rated.
Symptom Scale-8 (SSS-8) | Screening, treatment week 4 (post), and at the 3-month follow-up.
  Used to assess somatic symptoms and pain burden. SSS-8 consist of 8 items, each item is rated on a 5-point scale, with higher scores representing greater degree of pain problems. Self-rated.
Affective Control Scale, fear of anger subscale (ACS) | Screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up.
  Used to assess fear of anger. The fear of anger scale consists of 8 items, each rated on a 7-point scale, with higher scores indicating greater fear of anger.
State-Trait Anger Expression Inventory-2, Anger-Expression Out scale, and trait anger (STAXI-2; AX-O;T-ANG) | Screening, baseline week 4 (pre), treatment week 4 (post), and at the 3-month follow-up.
  Used to assess symptom severity of maladaptive expressions of anger and frequency of anger experiences (i.e., trait anger). The anger-expression out scale consists of 8 items, each rated on a 4-point scale with higher scores indicating greater problems with anger expression. The trait anger scale consists of 10 items, each rated on a 4-points scale, with higher scores indicating greater frequency of anger experiences. Self-rated.

OTHER OUTCOMES:
Demographic information | Screening
  For this study we collected information about the following: telephone number, e-mail, date of birth, gender, country of origin, partnership, living conditions (e.g., living alone, with children, and family), suspected of violent crime, convicted for violent crime, neuropsychiatric disorder (yes/no), highest education, employment, sick-leave, prior psychological treatment, current psychological treatment, and psychotropic medication.
Mini International Neuropsychiatric Interview (MINI | Screening
  A semi-structured interview used to assess psychiatric diagnoses during the screening process. Covers 17 of the most common psychiatric disorders in the Diagnostic Manual for Mental disorders - version 5 (DSM-5). Clinician-rated.
Risk for Violence Interview (RVI) | Screening
  A semi-structured interview, created by our research team, was used to screen for physical and psychological violence and abuse, both from a perpetrator- and victimization perspective. RVI builds upon the Revised Conflict Tactics Scale (CTS), and the Multidimensional Measure of Emotional Abuse (MMEA). Clinician-rated.
Treatment Credibility Scale (TCS) | Treatment week 2
  Used to assess treatment credibility. The scale consists of 6 items either rated on a 9-point scale or a percentage bar, with 10 % intervals (0-100 %). Higher scores indicate greater treatment credibility. Self-rated.
Client Satisfaction Questionnaire -8 (CSQ-8) | Treatment week 4 (post)
  Used to assess client satisfaction with treatment. This scale has 8 items, each rated on a 4-point scale, with higher scores indicating greater treatment satisfaction. Self-rated.
Questionnaire on adverse events experienced during internet-therapy | Treatment week 4 (post), and at 3-month follow-up.
  Used to assess adverse events related to treatment. In addition to being asked to report any negative or adverse during treatment, participants also got to answer this questionnaire. This questionnaire consists of 13 items representing potential adverse events that can be experienced during internet-treatment. Participants are asked to report the extent of impact of these events on their well-being using a 4-point scale, with higher scores indicating a greater impact. Self-rated.
Patient adherence | Treatment week 1-4
  Patient adherence will be monitored throughout the treatment by assessing completed treatment modules, completed exercises, completed homework, logged communication with the assigned therapist and time logged in on the treatment platform.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Hesser, Phd, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be publicly available according to national (Swedish) and European Union legislation and thus cannot be published in an open repository. However, if granted by the ethical review board in Stockholm, Sweden, aggregated data could be made available upon request.

REFERENCES:
- [Background] Bjureberg J, Ojala O, Berg A, Edvardsson E, Kolbeinsson O, Molander O, Morin E, Nordgren L, Palme K, Sarnholm J, Wedin L, Ruck C, Gross JJ, Hesser H. Targeting maladaptive anger with brief therapist-supported internet-delivered emotion regulation treatments: A randomized controlled trial. J Consult Clin Psychol. 2023 May;91(5):254-266. doi: 10.1037/ccp0000769. Epub 2022 Nov 21. PMID 36409100
- [Background] Burns JW, Quartana PJ, Bruehl S. Anger inhibition and pain: conceptualizations, evidence and new directions. J Behav Med. 2008 Jun;31(3):259-79. doi: 10.1007/s10865-008-9154-7. Epub 2008 May 23. PMID 18498056
- [Derived] Larsson J, Ojala O, Bjureberg J, Sederstrom P, Hvass O, Bjork P, Lidskog S, Hesser H. Online emotion regulation treatment for maladaptive anger inhibition - an open-label pilot with a pooled interrupted time series design. Cogn Behav Ther. 2025 Aug 4:1-16. doi: 10.1080/16506073.2025.2542355. Online ahead of print. PMID 40757961